CLINICAL TRIAL: NCT01316510
Title: Probiotics in Infants With Gastroschisis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 201018539
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2017-10

CONDITIONS: Gastroschisis
Keywords: Probiotic; bifidobacteria; intestinal motility
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifidobacteria infantis (Active Comparator): 1 billion organisms twice daily either through a feeding tube or by mouth for 6 weeks or until discharge (whichever happens first)
  Interventions: Dietary Supplement: Bifidobacteria infantis
- Placebo (Placebo Comparator): A dilute formulation of the elemental formula Nutramigen (diluted to look like the probiotic arm).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacteria infantis — 1 billion organisms twice daily either through a feeding tube or by mouth for 6 weeks or until discharge
  Arms: Bifidobacteria infantis
Other: Placebo — Dilute Nutramigen formula
  Arms: Placebo

SUMMARY:
Infants born with gastroschisis usually require surgery shortly after birth. After surgery the intestine is often unable to digest human milk or formula for weeks or months. During this time the baby has to remain in the hospital to receive special nutrition through an IV. How bacteria colonize the intestine in these babies is unknown. Probiotics are bacteria that appear to have beneficial effects on digestion. This study will test whether giving probiotic bacteria to babies after surgery for gastroschisis will change the bacteria in the intestine to be more like those of a healthy breast-fed baby.

DETAILED DESCRIPTION:
Infants with gastroschisis have decreased intestinal motility. This decrease in intestinal motility delays the introduction and advancement of feeds which prolongs hospitalization. The use of probiotic bacteria may improve intestinal motility. It is unknown whether the intestinal microbiota of infants with gastroschisis differs from that of healthy infants without gastroschisis and whether probiotics will change the microbiota. The primary outcome in this study is the composition of the fecal microbiota in infants with gastroschisis following surgical correction treated with Bifidobacterium infantis or placebo. We will also look at differences in hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Gastroschisis
* Born at or transferred to UC Davis Children's hospital

Exclusion Criteria:

* None

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Underwood, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Children's Hospital, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Powell WT, Borghese RA, Kalanetra KM, Mirmiran M, Mills DA, Underwood MA. Probiotic Administration in Infants With Gastroschisis: A Pilot Randomized Placebo-Controlled Trial. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):852-857. doi: 10.1097/MPG.0000000000001031. PMID 26545203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants were eligible for the study if they had confirmed gastroschisis at birth and gestational age at birth > 34 weeks. Parents were approached prior to or after the birth. All infants enrolled were inpatients in the NICU at UC Davis Children's Hospital in Sacramento CA. Enrollment began in March 2011 and was completed in Feb 2015.
Groups:
- Bifidobacterium Infantis: 1 billion organisms twice daily either through a feeding tube or by mouth for 6 weeks or until discharge (whichever happens first)
  Bifidobacterium infantis: 1 billion organisms twice daily either through a feeding tube or by mouth for 6 weeks or until discharge
Period: Overall Study
Arm/Group | Bifidobacterium Infantis | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bifidobacterium Infantis | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Customized [Median (Inter-Quartile Range); unit: Weeks]
  Gestational Age | 36.5 [35.75 to 37] | 37 [36 to 37] | 37 [36 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Birth weight [Mean (Standard Deviation); unit: Grams] | 2533 (431) | 2550 (342) | 2541 (380)

OUTCOME MEASURES:

1. Primary Outcome: Composition of the Fecal Microbiota
Description: Stools will be collected from messy diapers.
  Percentage bifidobacteria = total bifidobacteria per Group divided by the total bacteria per Group multiplied by 100% Percentage clostridia = total clostridia per Group divided by the total bacteria per Group multiplied by 100%
Time Frame: Final stool sample at 6 weeks
Population: Final stool sample
Measure: Number; unit: percentage of total bacteria
Arm/Group | Bifidobacterium Infantis | Placebo
Number analyzed (Participants) | 10 | 11
percentage of total bacteria
  Percentage bifidobacteria | 42 | 12
  Percentage clostridia | 1.1 | 14
Statistical Analysis 1: Comparison: Bifidobacterium Infantis vs Placebo; Primary outcome (percentage of bifidobacteria in the final stool specimen); Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Length of Hospital Stay
Description: Number of days from surgery until discharge
Time Frame: Initial discharge from the hospital
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bifidobacterium Infantis | Placebo
Number analyzed (Participants) | 12 | 12
days | 32.7 (11.1) | 43.6 (46.5)
Statistical Analysis 1: Comparison: Bifidobacterium Infantis vs Placebo; Secondary outcome (length of hospital stay) for all 24 infants (this included two infants with intestinal atresia, both in the placebo group); Test type: Superiority or Other; p = 0.44, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Bifidobacterium Infantis | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes